CLINICAL TRIAL: NCT01996865
Title: A Phase 3B Randomized Study of Lenalidomide (CC-5013) Plus Rituximab Maintenance Therapy Followed by Lenalidomide Single-Agent Maintenance Versus Rituximab Maintenance in Subjects With Relapsed/Refractory Follicular, Marginal Zone, or Mantle Cell Lymphoma
Brief Title: Lenalidomide Plus Rituximab Followed by Lenalidomide Versus Rituximab Maintenance for Relapsed/Refractory Follicular, Marginal Zone or Mantle Cell Lymphoma.
Acronym: MAGNIFY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-NHL-008
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Lymphoma, Mantle cell Lymphoma, Follicular Lymphoma, Marginal zone Lymphoma, Lenalidomide treatment, rituximab treatment, Non Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Lenalidomide + rituximab followed by lenalidomide (Experimental): Induction Period (12 cycles): Lenalidomide 20mg (10 mg if creatinine clearance ≥ 30 mL/min but < 60mL/min) by mouth (PO) daily (QD) on Days 1 to 21 of every 28-day cycle during cycles 1 through 12 and rituximab 375mg/m^2 intraveneously (IV) every week in Cycle 1 on Days 1, 8, 15, and 22 and on Day 1 of every 28-day cycle during cycles 3, 5, 7, 9, and 11, followed by a Maintenance Period (lasting 18 Cycles) that includes Lenalidomide 10 mg PO QD on Days 1 to 21 of every 28-day cycle during cycles 13 to 30 and rituximab 375 mg/m^2 IV on Day 1 of every 28-day cycle during cycles 13, 15, 17, 19, 21, 23, 25, 27, and 29 followed by an optional Maintenance Period (up to Progressive Disease) receiving Lenalidomide 10mg PO QD on Days 1 through 21 of every 28 day cycle until the disease progresses
  Interventions: Drug: Lenalidomide; Drug: Rituximab
- Arm B: Lenalidomide + rituximab followed by rituximab (Active Comparator): Induction Period (12 Cycles): Lenalidomide 20 mg PO QD (10 mg if creatinine clearance ≥ 30 mL/min but < 60 mL/min) on Days 1 to 21 of every 28-day cycle during cycles 1 to 12 and rituximab 375 mg/m^2 IV every week in cycle 1 on Days 1, 8, 15, and 22 and on Day 1 of every 28-day cycle during cycles 3, 5, 7, 9, and 11, followed by a Maintenance Period for 18 Cycles that includes: Rituximab 375 mg/m^2 IV on Day 1 of every 28-day cycle during cycles 13, 15, 17, 19, 21, 23, 25, 27, and 29
  Interventions: Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: CC-5013, Revlimid
Drug: Rituximab
  Other Names: Rituxan

SUMMARY:
Follicular lymphoma (FL), marginal zone lymphoma (MZL), and mantle cell lymphoma (MCL) are distinct histologic types of B-cell NHL. Lenalidomide is an immunomodulatory agent with direct and immune-mediated mechanisms of action, as well as clinical activity in NHL. Recent studies in frontline and relapsed/refractory NHL show high activity for lenalidomide plus rituximab (R2), supporting further study of this combination.

DETAILED DESCRIPTION:
MAGNIFY (NCT01996865) is a phase 3b, multicenter, open-label study of patients with grades 1-3b or transformed follicular lymphoma (FL), marginal zone lymphoma (MZL), or mantle cell lymphoma (MCL) who received ≥1 prior therapy and had stage I-IV, measurable disease. ~500 patients are planned for enrollment in 12 cycles of R2 induction, with a projected ~314 patients with ≥SD after induction randomized (1:1) to two maintenance arms. Induction includes oral lenalidomide 20 mg/day, days 1-21 per 28-day cycle (d1-21/28) plus IV rituximab 375 mg/m2, days 1, 8, 15, and 22 of cycle 1 and day 1 of cycles 3, 5, 7, 9, and 11 (28-day cycles). Patients are then randomized to maintenance lenalidomide 10 mg/day, d1-21/28, cycles 13-30, plus rituximab 375 mg/m2, day 1 of cycles 13, 15, 17, 19, 21, 23, 25, 27, and 29 (R2, Arm A), or rituximab alone (same schedule, Arm B). Patients receiving R2 maintenance after 18 cycles may continue maintenance lenalidomide monotherapy 10 mg/day, d1-21/28 (per patient and/or investigator discretion), until disease progression as tolerated. The primary endpoint is progression-free survival (per modified 1999 IWG criteria). Secondary endpoints include safety, overall survival, response rates, duration of response, and quality of life (exploratory). Patients will be followed for ≥5 years after the last patient initiated induction therapy. Enrollment in MAGNIFY began in March 2014; as of Jan 2016, 133 patients are enrolled.

ELIGIBILITY:
Inclusion Criteria:

-- Age ≥18 years

* Histologically confirmed Follicular Lymphoma (FL, Grade 1, 2, 3a, or 3b), Transformed FL, Marginal Zone Lymphoma, or Mantle Cell Lymphoma
* Must have documented relapsed, refractory or Progressive Disease after last treatment with systemic therapy
* Bi-dimensionally measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance status < 2
* Adequate bone marrow function
* Willingness to follow pregnancy precautions

Exclusion Criteria:

* Histology other than follicular or marginal zone lymphoma or clinical evidence of transformation or Grade 3b follicular lymphoma
* Any medical condition (other than the underlying lymphoma) that requires chronic steroid use
* Subjects taking corticosteroids during the last 1 week prior treatment, unless administered at a dose equivalent to < 20 mg/day of prednisone
* Systemic anti-lymphoma therapy within 28 days or use of antibody agents within 4 weeks use of radioimmunotherapy within 3 months
* Known seropositive for or active viral infection with hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV)
* Known sensitivity or allergy to murine products
* Presence or history of central nervous system involvement by lymphoma. Subjects who are at a risk for a thromboembolic event and are not willing to take prophylaxis for it
* Any condition that places the subject at unacceptable risk if he/she were to participate in the study or that confounds the ability to interpret data from the study

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (126):
- United States (110):
  - Local Institution - 055, Tucson, Arizona
  - Local Institution - 077, Little Rock, Arkansas
  - Local Institution - 079, Berkeley, California
  - Local Institution - 142, Concord, California
  - Bay Area Cancer Research Group, LLC, Pleasant Hill, California
  - Sutter Hematology and Oncology, Sacramento, California
  - Local Institution - 032, San Diego, California
  - Local Institution - 130, Santa Barbara, California
  - Local Institution - 052, Boulder, Colorado
  - Local Institution - 106, Denver, Colorado
  - Colorado Cancer Research Program, Denver, Colorado
  - Local Institution - 062, Glenwood Springs, Colorado
  - Praxair Cancer Center Danbury, Danbury, Connecticut
  - Medical Oncology and Blood Disorders, LLP, Manchester, Connecticut
  - Local Institution - 041, Norwalk, Connecticut
  - Hematology Oncology Associates, PC, Stamford, Connecticut
  - Local Institution - 149, Trumbull, Connecticut
  - Local Institution - 116, Waterbury, Connecticut
  - Local Institution - 068, Fleming Island, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Local Institution - 054, Ocala, Florida
  - Local Institution - 114, Pensacola, Florida
  - Local Institution - 011, Marietta, Georgia
  - Local Institution - 083, Newnan, Georgia
  - Local Institution - 108, Elk Grove Village, Illinois
  - United States Department of Veterans Affairs - VA Great Lakes Health Care System - Edward Hines Jr, Hines, Illinois
  - Local Institution - 159, Hinsdale, Illinois
  - Local Institution - 056, Niles, Illinois
  - Local Institution - 028, Park Ridge, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - American Health Network of Indiana, LLC, New Albany, Indiana
  - McFarland Clinic, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - Local Institution - 019, Fairway, Kansas
  - Local Institution - 350, Great Bend, Kansas
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Local Institution - 138, Louisville, Kentucky
  - Local Institution - 143, Waterville, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Local Institution - 030, Baltimore, Maryland
  - Associates Of Oncology/Hematology, P.C., Rockville, Maryland
  - Local Institution - 051, Ann Arbor, Michigan
  - Local Institution - 033, Lansing, Michigan
  - Local Institution - 164, Rochester, Minnesota
  - Local Institution - 050, Bolivar, Missouri
  - Local Institution - 103, Columbia, Missouri
  - Local Institution - 013, Springfield, Missouri
  - Local Institution - 042, St Louis, Missouri
  - Local Institution - 003, Lincoln, Nebraska
  - Local Institution - 098, Lebanon, New Hampshire
  - Summit Medical Group Overlook Oncology Center, Berkeley Heights, New Jersey
  - Veterans Affairs New Jersey Health Care System, East Orange, New Jersey
  - Local Institution - 080, Englewood, New Jersey
  - Local Institution - 025, Mount Holly, New Jersey
  - Saint Peter'S University Hospital, New Brunswick, New Jersey
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - C.R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Broome Oncology, LLC, Johnson City, New York
  - Local Institution - 152, Lake Success, New York
  - Local Institution - 023, Kinston, North Carolina
  - Local Institution - 039, Raleigh, North Carolina
  - Summa Health System Akron City Hospital Laboratory, Akron, Ohio
  - Aultman Hospital, Canton, Ohio
  - Local Institution - 161, Cincinnati, Ohio
  - Local Institution - 047, Cleveland, Ohio
  - Local Institution - 045, Columbus, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Local Institution - 037, Oklahoma City, Oklahoma
  - Local Institution - 059, Eugene, Oregon
  - Hematology Oncology Associates, P.C., Medford, Oregon
  - Local Institution - 073, Greenville, South Carolina
  - Spartanburg Regional Healthcare System - Gibbs Cancer Center & Research Institute, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Local Institution - 153, Sioux Falls, South Dakota
  - Baptist Cancer Center, Memphis, Tennessee
  - Local Institution - 076, Memphis, Tennessee
  - Local Institution - 166, Amarillo, Texas
  - Arlington Cancer Center, Arlington, Texas
  - Texas Oncology-Arlington South, Arlington, Texas
  - Local Institution - 105, Dallas, Texas
  - Local Institution - 026, Houston, Texas
  - Local Institution - 067, Houston, Texas
  - Local Institution - 008, Houston, Texas
  - Local Institution - 021, Plano, Texas
  - Local Institution - 071, Round Rock, Texas
  - Local Institution - 070, San Antonio, Texas
  - Local Institution - 058, San Antonio, Texas
  - Local Institution - 111, Temple, Texas
  - Local Institution - 094, Tyler, Texas
  - Local Institution - 163, Tyler, Texas
  - Local Institution - 057, Webster, Texas
  - Local Institution - 090, Salt Lake City, Utah
  - Rutland Regional Medical Center, Rutland, Vermont
  - Local Institution - 053, Christiansburg, Virginia
  - Local Institution - 129, Fort Belvoir, Virginia
  - Local Institution - 081, Norfolk, Virginia
  - Cancer Treatment Center of America, Portsmouth, Virginia
  - PeaceHealth St. Joseph Medical Center, Bellingham, Washington
  - Local Institution - 049, Gig Harbor, Washington
  - Local Institution - 119, Olympia, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Local Institution - 104, Vancouver, Washington
  - Local Institution - 099, Walla Walla, Washington
  - Local Institution - 006, Wenatchee, Washington
  - Local Institution - 038, Morgantown, West Virginia
  - Aurora Health Care Aurora Research, Milwaukee, Wisconsin
  - Local Institution - 301, Mukwonago, Wisconsin
  - Local Institution - 300, Oconomowoc, Wisconsin
  - Local Institution - 101, Waukesha, Wisconsin
- Germany (15):
  - Local Institution - 208, Berlin
  - Local Institution - 202, Bremen
  - Local Institution - 213, Cologne
  - Local Institution - 205, Frankfurt
  - Local Institution - 211, Frechen
  - Local Institution - 200, Giessen
  - Local Institution - 203, Hanover
  - Local Institution - 206, Kassel
  - Local Institution - 210, Marburg
  - Local Institution - 215, Mönchengladbach
  - Local Institution - 204, München
  - Local Institution - 212, Münster
  - Local Institution - 201, Potsdam
  - Local Institution - 207, Ravensberg
  - Local Institution - 209, Würzburg
- Local Institution - 029, San Juan, Puerto Rico

REFERENCES:
- [Background] Leonard JP, Trneny M, Izutsu K, Fowler NH, Hong X, Zhu J, Zhang H, Offner F, Scheliga A, Nowakowski GS, Pinto A, Re F, Fogliatto LM, Scheinberg P, Flinn IW, Moreira C, Cabecadas J, Liu D, Kalambakas S, Fustier P, Wu C, Gribben JG; AUGMENT Trial Investigators. AUGMENT: A Phase III Study of Lenalidomide Plus Rituximab Versus Placebo Plus Rituximab in Relapsed or Refractory Indolent Lymphoma. J Clin Oncol. 2019 May 10;37(14):1188-1199. doi: 10.1200/JCO.19.00010. Epub 2019 Mar 21. PMID 30897038
- [Background] Becnel MR, Nastoupil LJ, Samaniego F, Davis RE, You MJ, Green M, Hagemeister FB, Fanale MA, Fayad LE, Westin JR, Wang M, Oki Y, Forbes SG, Feng L, Neelapu SS, Fowler NH. Lenalidomide plus rituximab (R2 ) in previously untreated marginal zone lymphoma: subgroup analysis and long-term follow-up of an open-label phase 2 trial. Br J Haematol. 2019 Jun;185(5):874-882. doi: 10.1111/bjh.15843. Epub 2019 Mar 28. PMID 30919940
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 503 participants joined this study. All participants started in the induction period; only those who did not progress after 12 cycles of treatment were randomized to receive treatment in the maintenance period.
Groups:
- Induction Period: Lenalidomide + Rituximab: Induction Period (12 cycles): participants received lenalidomide 20 mg (10 mg if creatinine clearance ≥ 30 mL/min but < 60 mL/min) once daily on Days 1 to 21 of every 28-day Cycle for Cycles 1 to 12 AND rituximab 375 mg/m2 every week in Cycle 1 (Days 1, 8, 15, and 22) and Day 1 of every 28-day Cycle for Cycles 3, 5, 7, 9, and 11
- Arm A: Lenalidomide + Rituximab: Maintenance Period (18 Cycles): lenalidomide 10 mg once daily on Days 1 to 21 of every 28-day Cycle for Cycles 13 to 30 AND rituximab 375 mg/m2 on Day 1 of every 28-day Cycle for Cycles 13, 15, 17, 19, 21, 23, 25, 27, and 29. Followed by Optional Maintenance Period (up to PD): Lenalidomide 10 mg once daily on Days 1 to 21 of every 28-day Cycle up to PD. This treatment will be at the discretion of the participant and the investigator.
- Arm B: Rituximab: Maintenance Period (18 Cycles): participants received rituximab 375 mg/m2 on Day 1 of every 28-day Cycle for Cycles 13, 15, 17, 19, 21, 23, 25, 27, and 29
Period: Induction Period
Arm/Group | Induction Period: Lenalidomide + Rituximab | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Started (Randomized) | 503 | 0 | 0
Treated | 500 | 0 | 0
Completed | 284 | 0 | 0
Not Completed | 219 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Progressive Disease | 4 | 0 | 0
Not completed — Lost to Follow-up | 10 | 0 | 0
Not completed — Other Reasons | 13 | 0 | 0
Not completed — Adverse Event | 20 | 0 | 0
Not completed — Withdrawal by Subject | 60 | 0 | 0
Not completed — Death | 111 | 0 | 0
Period: Maintenance Period
Arm/Group | Induction Period: Lenalidomide + Rituximab | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Started (Randomized) | 0 | 135 | 132
Treated | 0 | 134 | 132
Completed | 0 | 78 | 89
Not Completed | 0 | 57 | 43
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Other reasons | 0 | 8 | 5
Not completed — Progressive Disease | 0 | 6 | 23
Not completed — Withdrawal by Subject | 0 | 18 | 4
Not completed — Adverse Event | 0 | 7 | 7
Not completed — Death | 0 | 15 | 3
Not completed — Lost to Follow-up | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants started in the induction and maintenance periods and are accounted for in this arm.
Groups:
- Overall Study: All participants who were enrolled into the study.
Arm/Group | Overall Study
Number analyzed (Participants) | 503
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 209
  >=65 years | 294
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215
  Male | 288
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33
  Not Hispanic or Latino | 463
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 17
  White | 468
  More than one race | 0
  Unknown or Not Reported | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time from the date of first dose of maintenance therapy to the date of the first objective documentation of tumor progression or death due to any cause. Analysis was based on Kaplan Meier estimates. The PFS events were determined using a modification of the IWG 1999 criteria.
Time Frame: From the first dose date of maintenance therapy to objective disease progression or death from any cause, whichever occurs first (up to approximately 432 weeks)
Population: All randomized participants in Arm A and Arm B, as prespecified in the protocol
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 135 | 132
Weeks | 263.1 [166.1 to NA] — Upper limit not calculated due to insufficient number of events. | 229.1 [173.7 to NA] — Upper limit not calculated due to insufficient number of events.
Statistical Analysis 1: Comparison: Arm A: Lenalidomide + Rituximab vs Arm B: Rituximab; Test type: Other; p = 0.3296, Regression, Cox; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.6 to 1.2]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time between the first dose date of maintenance therapy and death from any cause. Participants who complete the study and are still alive at the time of the clinical data cutoff date will be censored at the last visit date or the last contact date, whichever is later. Participants who were lost to follow-up prior to the clinical data cut-off date will also be censored at the time of the last contact. Analysis was based on Kaplan Meier estimates and Hazard Ratio (HR).
Time Frame: From the first dose date of maintenance therapy to death from any cause (up to approximately 480 weeks)
Population: All randomized participants in Arm A and Arm B, as prespecified in the protocol
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 135 | 132
Weeks | NA [439.4 to NA] — Median and upper limit not calculated due to insufficient number of events. | NA [395.7 to NA] — Median and upper limit not calculated due to insufficient number of events.
Statistical Analysis 1: Comparison: Arm A: Lenalidomide + Rituximab vs Arm B: Rituximab; Test type: Other; p = 0.1222, Regression, Cox; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.4 to 1.1]

3. Secondary Outcome: Improvement of Response (IOR)
Description: Improvement of Response (IOR) is the percentage of participants with improved tumor response during the maintenance phase (converted from partial response at end of induction to complete response or complete response unconfirmed as best response) and participants who converted from stable disease at the end of induction period to partial response or better as best response during maintenance phase.
Time Frame: From the first dose date of maintenance therapy to death from any cause (up to approximately 432 weeks)
Population: All randomized participants in Arm A and Arm B, as prespecified in the protocol
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 135 | 132
Percentage of participants | 20 [13.6 to 27.7] | 11.4 [6.5 to 18.0]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: The overall response rate (ORR) is defined as the percentage of participants with a best response of at least partial response (including complete response, complete response unconfirmed and partial response) after the first dose date of maintenance therapy and prior to any treatment change.
Time Frame: From the first dose date of maintenance therapy up to CR, CRu, PR, or treatment change (up to approximately 432 weeks)
Population: All randomized participants in Arm A and Arm B, as prespecified in the protocol
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 115 | 105
Percentage of participants | 85.2 [78.1 to 90.7] | 79.5 [71.7 to 86.1]

5. Secondary Outcome: Complete Response Rate (CRR)
Description: Best Complete Response Rate (CRR), defined as the proportion of participants with a best response of at least CRu (including CR and CRu) after the first dose date of maintenance therapy and prior to any treatment change.
Time Frame: From the first dose date of maintenance therapy up to CR or CRu (up to approximately 432 weeks)
Population: All randomized participants in Arm A and Arm B, as prespecified in the protocol
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 135 | 132
Percentage of participants | 60.7 [52.0 to 69.0] | 58.3 [49.4 to 66.8]

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR is from initial response (at least CRu) after the first dose date of maintenance therapy and prior to treatment change to documented disease progression or death. Participants who have not progressed or died at the time of the clinical data cutoff date will be censored at the last assessment showing no progression. Participants who change treatment without evidence of disease progression will be censored at the last assessment showing no progression prior to treatment change. Analysis was based on Kaplan Meier estimates.
Time Frame: From the initial response (at least PR) after the first dose date of maintenance therapy and prior to treatment change to documented disease progression or death, whichever occurs first (up to approximately 432 weeks)
Population: The analysis is only performed for participants who have achieved PR or better after the first dose date of maintenance therapy and prior to any treatment change.
  Arm B includes 3 additional participants who achieved CR/CRu/PR in the follow-up period.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 115 | 108
Weeks | 268.3 [168.0 to NA] — Upper limit not calculated due to insufficient number of events | 306.0 [183.7 to NA] — Upper limit not calculated due to insufficient number of events

7. Secondary Outcome: Time to Next Anti-lymphoma Treatment
Description: Time to next anti-lymphoma treatment is defined as the time from the first dose date of maintenance therapy to the time of first documented administration of new anti-lymphoma therapy. Participants without new treatment therapy will be censored at the last visit. Analysis was based on Kaplan Meier estimates.
Time Frame: From the first dose date of maintenance therapy to the time of first documented administration of new anti-lymphoma therapy (up to approximately 300 weeks)
Population: All randomized participants in Arm A and Arm B, as prespecified in the protocol
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 135 | 132
Weeks | NA [300.4 to NA] — Median and upper limit not calculated due to insufficient number of events | NA [283.4 to NA] — Median and upper limit not calculated due to insufficient number of events

8. Secondary Outcome: Time to Histological Transformation
Description: Time to histological transformation is defined as from the first dose date of maintenance therapy to the time of histological transformation as measured based on documentation of histological transformation (as assessed by the investigator). Analysis was based on Kaplan Meier estimates.
  In case of clinical suspicion of transformation, including rapid disease progression, unexpected changes in "B" symptoms or rapidly increasing LDH, a biopsy should be performed. In this clinical trial, histological transformation will be considered disease progression. This endpoint will not be calculated for participants randomized with transformed Follicular Lymphoma (tFL).
Time Frame: From the first dose date of maintenance therapy to the time of histological transformation (up to approximately 432 weeks)
Population: All randomized participants in Arm A and Arm B without transformed Follicular Lymphoma (tFL)
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 133 | 129
Weeks | NA [NA to NA] — Median, lower and upper limit not calculated due to insufficient number of events. | NA [NA to NA] — Median, lower and upper limit not calculated due to insufficient number of events.

9. Secondary Outcome: Duration of Complete Response (DOCR)
Description: Duration of complete response (DOCR) is calculated as the time from the initial response (CR or CRu) after the first dose date of maintenance therapy and prior to treatment change to documented disease progression or death. Analysis was based on Kaplan Meier estimates. Participants who have not progressed or died at the time of the clinical data cutoff date will be censored at the last assessment showing no progression. Participants who change treatment without evidence of disease progression will be censored at the last assessment showing no progression prior to treatment change.
Time Frame: From the initial CR/CRu after the first dose date of maintenance therapy and prior to treatment change to documented disease progression or death, whichever occurs first (up to approximately 432 weeks)
Population: The analysis is only performed for participants who have achieved CR or CRu after the first dose date of maintenance therapy and prior to any treatment change.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 85 | 82
Weeks | 298.0 [176.0 to NA] — Upper limit not calculated due to insufficient number of events | NA [221.1 to NA] — Median and upper limit not calculated due to insufficient number of events

10. Secondary Outcome: Participants Experiencing Treatment Emergent Adverse Events (TEAEs)
Description: Number of participants experiencing AEs, SAEs, AEs leading to study discontinuation, and AEs of interest (AEIs). An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. SAEs is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization; results significant disability; or is a congenital anomaly/birth defect. TEAEs are defined as AEs with an onset date on or after the first dose of study treatment up to 30 days after the last dose of study treatment in the study, or if a pre-existing condition worsens in severity or becomes serious after receiving the first dose of study treatment.
Time Frame: From first dose up to 30 days after last dose (up to approximately 64 weeks for induction period and 427 weeks for maintenance period)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Lenalidomide + Rituximab | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 500 | 134 | 132
Participants
  Participants experiencing at least one TEAE | 499 | 133 | 120
  Participants experiencing at least one serious TEAE | 172 | 57 | 22

11. Secondary Outcome: Participants Experiencing Adverse Events Related to Vital Signs
Description: The number of participants who experienced adverse events related to vital sign measurements
Time Frame: as for outcome 10
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Lenalidomide + Rituximab | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 500 | 134 | 132
Participants
  Hypertension | 34 | 9 | 6
  Hypotension | 22 | 4 | 5
  Hypoxia | 5 | 2 | 0

12. Secondary Outcome: Participants With Grade 3 or Grade 4 Hematology Parameters
Description: Clinical laboratory values in induction period include any laboratory values that are taken after the first dose date of induction therapy through 28 days after the last dose date of induction therapy or before the first dose date of maintenance therapy, whichever is earlier. Graded according to the NCI CTCAE version 4.03, except for tumor flare reaction, which is accessed using NCI CTCAE version 3.0. Participants with zero maximum grade are excluded.
Time Frame: as for outcome 10
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Lenalidomide + Rituximab | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 500 | 134 | 132
Participants
  Anemia - Grade 3 | 31 | 7 | 0
  Leukopenia - Grade 3 | 101 | 19 | 6
  Thrombocytopenia - Grade 3 | 29 | 2 | 1
  Neutropenia - Grade 3 | 103 | 24 | 10
  Lymphopenia - Grade 3 | 126 | 31 | 21
  Anemia - Grade 4 | 0 | 0 | 0
  Leukopenia - Grade 4 | 17 | 5 | 0
  Thrombocytopenia - Grade 4 | 7 | 0 | 0
  Neutropenia - Grade 4 | 94 | 25 | 6
  Lymphopenia - Grade 4 | 20 | 10 | 2

13. Secondary Outcome: Participants With Grade 3 or Grade 4 Serum Chemistry Parameters
Description: Clinical laboratory values in induction period include any laboratory values that are taken after the first dose date of induction therapy through 28 days after the last dose date of therapy. Graded according to the NCI CTCAE version 4.03, except for tumor flare reaction, which is accessed using NCI CTCAE version 3.0. Participants with zero maximum grade are excluded.
Time Frame: as for outcome 10
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Lenalidomide + Rituximab | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
Number analyzed (Participants) | 500 | 134 | 132
Participants
  Hypokalemia - Grade 3 | 30 | 8 | 4
  Hyperkalemia- Grade 3 | 4 | 0 | 1
  Hypocalcemia - Grade 3 | 7 | 1 | 0
  Hypercalcemia - Grade 3 | 7 | 0 | 0
  Hypophosphatemia - Grade 3 | 17 | 6 | 2
  Hypercreatininemia - Grade 3 | 3 | 1 | 0
  Hyperuricemia - Grade 3 | 40 | 13 | 20
  Alanine Aminotransferase Increased - Grade 3 | 14 | 3 | 0
  Aspartate Aminotransferase Increased - Grade 3 | 9 | 1 | 0
  Hyperbilirubinemia - Grade 3 | 5 | 3 | 1
  Hypokalemia - Grade 4 | 4 | 0 | 0
  Hyperkalemia- Grade 4 | 1 | 2 | 0
  Hypocalcemia - Grade 4 | 5 | 5 | 2
  Hypercalcemia - Grade 4 | 3 | 5 | 0
  Hypophosphatemia - Grade 4 | 1 | 1 | 1
  Hypercreatininemia - Grade 4 | 1 | 2 | 0
  Hyperuricemia - Grade 4 | 9 | 4 | 0
  Alanine Aminotransferase Increased - Grade 4 | 0 | 0 | 0
  Aspartate Aminotransferase Increased - Grade 4 | 0 | 0 | 0
  Hyperbilirubinemia - Grade 4 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose of study treatment to study completion, (up to approximately 10 years). SAEs and Other AEs were assessed from first dose to 30 days following last dose (up to approximately 64 weeks for induction period and 427 weeks for maintenance period).
Arm/Group | Induction Period: Lenalidomide + Rituximab | Arm A: Lenalidomide + Rituximab | Arm B: Rituximab
All-Cause Mortality (participants affected / at risk) | 112/500 | 26/134 | 32/132
Serious Adverse Events (participants affected / at risk) | 172/500 | 57/134 | 22/132
Other Adverse Events (participants affected / at risk) | 491/500 | 129/134 | 106/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Period: Lenalidomide + Rituximab (N=500) | Arm A: Lenalidomide + Rituximab (N=134) | Arm B: Rituximab (N=132)
Pneumonia (Infections and infestations) | 18 | 8 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 10 | 5
Anaemia (Blood and lymphatic system disorders) | 8 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 15 | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 9 | 3 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Trifascicular block (Cardiac disorders) | 0 | 1 | 0
Ear canal stenosis (Ear and labyrinth disorders) | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 0
Colitis (Gastrointestinal disorders) | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Epiploic appendagitis (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0 | 1
Volvulus of small bowel (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Asthenia (General disorders) | 3 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 3 | 2
Sudden death (General disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic haematoma (Hepatobiliary disorders) | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Contrast media allergy (Immune system disorders) | 1 | 0 | 0
Contrast media reaction (Immune system disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 3 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 5 | 3 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 2 | 0 | 0
Coronavirus infection (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1
Disseminated varicella zoster virus infection (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Histoplasmosis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Joint abscess (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia aspiration (Infections and infestations) | 3 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 2 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0
Psoas abscess (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 7 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 3 | 0
Urosepsis (Infections and infestations) | 2 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 3 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 8 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 5 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Bell's palsy (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0
Transient global amnesia (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 1 | 0
Device occlusion (Product Issues) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Granulomatous pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Period: Lenalidomide + Rituximab (N=500) | Arm A: Lenalidomide + Rituximab (N=134) | Arm B: Rituximab (N=132)
Anaemia (Blood and lymphatic system disorders) | 77 | 12 | 8
Leukopenia (Blood and lymphatic system disorders) | 67 | 13 | 9
Lymphopenia (Blood and lymphatic system disorders) | 33 | 5 | 3
Neutropenia (Blood and lymphatic system disorders) | 217 | 54 | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 74 | 9 | 5
Tinnitus (Ear and labyrinth disorders) | 5 | 7 | 3
Hypothyroidism (Endocrine disorders) | 14 | 7 | 4
Vision blurred (Eye disorders) | 18 | 9 | 0
Abdominal pain (Gastrointestinal disorders) | 57 | 13 | 8
Constipation (Gastrointestinal disorders) | 146 | 12 | 2
Diarrhoea (Gastrointestinal disorders) | 176 | 56 | 11
Dry mouth (Gastrointestinal disorders) | 31 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 35 | 4 | 0
Nausea (Gastrointestinal disorders) | 150 | 15 | 6
Stomatitis (Gastrointestinal disorders) | 37 | 3 | 3
Vomiting (Gastrointestinal disorders) | 54 | 10 | 4
Chills (General disorders) | 43 | 5 | 5
Fatigue (General disorders) | 225 | 27 | 15
Influenza like illness (General disorders) | 14 | 7 | 1
Oedema peripheral (General disorders) | 81 | 14 | 3
Pyrexia (General disorders) | 50 | 14 | 5
Hypogammaglobulinaemia (Immune system disorders) | 8 | 7 | 2
Bronchitis (Infections and infestations) | 23 | 12 | 5
COVID-19 (Infections and infestations) | 0 | 8 | 0
Nasopharyngitis (Infections and infestations) | 26 | 5 | 3
Pneumonia (Infections and infestations) | 35 | 17 | 5
Sinusitis (Infections and infestations) | 43 | 16 | 11
Upper respiratory tract infection (Infections and infestations) | 65 | 22 | 14
Urinary tract infection (Infections and infestations) | 41 | 11 | 4
Fall (Injury, poisoning and procedural complications) | 24 | 13 | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 53 | 0 | 0
Alanine aminotransferase increased (Investigations) | 30 | 5 | 2
Aspartate aminotransferase increased (Investigations) | 22 | 7 | 4
Blood creatinine increased (Investigations) | 22 | 12 | 4
Lymphocyte count decreased (Investigations) | 11 | 7 | 3
Weight decreased (Investigations) | 34 | 14 | 4
White blood cell count decreased (Investigations) | 20 | 10 | 1
Decreased appetite (Metabolism and nutrition disorders) | 69 | 8 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 24 | 8 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 17 | 8 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 63 | 16 | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 27 | 6 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 68 | 23 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 57 | 9 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 64 | 11 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 31 | 8 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 25 | 10 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 | 11 | 9
Dizziness (Nervous system disorders) | 68 | 14 | 7
Dysgeusia (Nervous system disorders) | 30 | 3 | 0
Headache (Nervous system disorders) | 66 | 15 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 56 | 14 | 6
Anxiety (Psychiatric disorders) | 31 | 8 | 3
Insomnia (Psychiatric disorders) | 50 | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 103 | 41 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 73 | 18 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 23 | 10 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 37 | 9 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 19 | 7 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 21 | 10 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 41 | 4 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 39 | 8 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 96 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 33 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 82 | 6 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 30 | 6 | 2
Hypertension (Vascular disorders) | 34 | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT01996865/Prot_SAP_000.pdf